CLINICAL TRIAL: NCT02845245
Title: CIDUCT: Comminuted Intra-Articular Distal Tibia Fracture Fixation Using Computer Surgical Planning and 3D Prototyping Techniques
Brief Title: Comminuted Intra-Articular Distal Tibia Fracture Fixation Using Computer Techniques
Acronym: CIDUCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goal was not met.
Sponsor: Inova Health Care Services (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Robert A. Hymes, Orthopaedic surgeon, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-2256
Record Dates: First submitted 2016-05-26; First posted 2016-07-27 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Tibial Fractures
Keywords: Comminuted intra-articular distal tibia fractures; 3D printing; pre-operative planning
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of care imaging techniques (3D CT scan and plain film radiographs) will be obtained for the surgeon to pre-operatively plan the surgery.
  Interventions: Other: 3D CT scan; Other: Plain film radiographs
- Intervention (Experimental): A 3D printed plastic model prototype will be developed for the surgeon to use, in addition to the standard of care imaging techniques (3D CT scan and plain film radiographs), to pre-operatively plan the surgery.
  Interventions: Other: 3D printed plastic model prototype; Other: 3D CT scan; Other: Plain film radiographs

INTERVENTIONS:
Other: 3D printed plastic model prototype
  Arms: Intervention
Other: 3D CT scan
Other: Plain film radiographs

SUMMARY:
Comminuted intra-articular distal tibia fractures (OTA 43-C) typically are the result of high-energy trauma such as motor vehicle collisions or fall from a height. They are complex injuries often associated with significant fragment displacement and severe soft tissue injury, a combination that has long challenged orthopedic surgeons. Traditionally, surgeons use plain film (X-ray) and CT scans (2 or 3 dimensional) to determine fracture pattern and displacement. Yet, in some cases, it is still difficult to identify the relationship among bone fragments, which often makes articular restoration challenging. As a result, patients with non-anatomic joint reconstructions have a higher rate of poor outcomes.

The primary objective of this study will be to compare patient outcomes in two groups, one group who will receive enhanced pre-operative planning (3D printed plastic prototype + standard of care [SOC] imaging with 3D CT scan + plain film radiographs) and a second group who will receive pre-operative planning using SOC imaging alone (3D CT scan + plain film radiographs only). Patient outcomes collected throughout the 12 month post-operative period will include an assessment of radiographic fracture healing (union, non-union, malunion), pain using a Numeric Pain Rating Scale, Olerud and Molander Score based on patient's self-report, and development of complications (infection, wound healing, re-operation, and re-hospitalizations). The secondary objective of this study will be to evaluate whether utilizing an enhanced pre-operative plan with a 3D printed plastic prototype altered the original pre-operative plan based on SOC imaging alone (3D CT scan + plain film radiographs only).

DETAILED DESCRIPTION:
1. Recruitment Patients with a comminuted distal tibia fracture (OTA 43-C type) who present for care at Inova Fairfax Medical Campus (IFMC) or at the Inova Medical Group (IMG) Orthopaedic outpatient clinic will be eligible for consent and possible enrollment in this study. Patients will not be compensated for participating in this study. Given that this is a convenience sample of patients who present with an acute traumatic injury, there are no plans to advertise or recruit patients.
2. Subject Randomization and Blinding Procedures Eligible patients will be randomized in equal proportions to one of two groups (enhanced pre-operative planning vs. SOC pre-operative planning) using an electronic randomization system with a simple randomization table. After consent and inclusion/exclusion criteria have been confirmed, subjects will be randomized by a research coordinator/associate. All surgeons will be temporarily blinded to the randomization assignment, in order to complete an unbiased pre-operative plan (pre-randomization survey) using the SOC imaging alone (plain film radiographs and 3D CT scan). After the pre-operative plan (pre-randomization survey) is completed by the attending surgeon (using the SOC imaging alone) and submitted to the research coordinator/ associate, the surgeon will be informed of the randomization assignment. For subjects randomized to the enhanced pre-operative planning group, the surgeon will then be provided the 3D prototype and be asked to complete a post-randomization survey capturing their pre-operative plan. The biomechanics lab with arrange with the research coordinator/associate for delivery of the 3D prototype, ensuring that the temporary blinding of treatment assignment is not broken. A post-randomization survey will not be administered to surgeons with subjects randomized to the SOC group.

   Subjects will not be blinded to the assigned group. However, in order to ensure the temporary blind is maintained with the attending surgeon who will be performing the definitive surgery, the subject won't be informed of their randomization assignment until the time of definitive surgery.
3. Standard of Care Procedures Prior to Definitive Surgery: All Groups The following pre-operative care described is the standard of practice and is a general summary of the care that will be given to all study patients prior to their definitive surgery, regardless of treatment group assignment. There are two scenarios with which patients will be eligible and approached for participation in this study: 1). stable fracture treated with a splint, and 2). unstable (open or closed) fracture requiring external-fixator surgery.

   All patients will be initially evaluated in the emergency department (ED) by a member of the orthopaedic trauma team. Patients with an axially stable injury will undergo manual realignment and application of a well-padded posterior with U-shaped plaster splint. A computed tomography (CT) scanning with sagittal, coronal reconstructions and 3D reformations will be obtained in the ED; and then sent home after learning to crutch ambulate, with instructions for continued strict elevation, non-weight bearing, and follow-up in the clinic. Once these patients are seen in the clinic, it is determined that surgery is required and the patient is subsequently scheduled for definitive surgery, to occur after resolution of swelling and normalization of skin.

   Patients who present in the ED with axially unstable-closed fractures on initial plain radiographs will undergo closed reduction and be admitted to the hospital for surgical placement of a temporizing, spanning external-fixator (Depuy Synthes Inc. West Chester, PA). Patients with axially unstable-open fractures will be administered intravenous antibiotics and tetanus update on presentation to the ED, and will go to the operating room for urgent initial debridement and placement of a temporizing, spanning external-fixator. Patients with unstable fractures (open or closed) will have computed tomography (CT) scanning with sagittal, coronal reconstructions and 3D reformations after placement of an external-fixator. Patients will be discharged with appropriate placement (home vs. acute rehab vs. SNF) after evaluation by physical therapy and have their definitive surgery scheduled. All patients will be non-weight bearing to the study injury limb. Definitive operative fixation will occur after resolution of swelling and normalization of skin.
4. Study Procedures: Pre-operative Surgery Planning and open treatment and internal fixation (ORIF) Surgery

   4.1 Standard of Care In the control group, 20 patients will have standard of care treatment, which includes pre-operative evaluation and surgical planning based on plain films (3 views: anterior, lateral and oblique) and CT scans with sagittal, coronal and 3D reformations. Operative fixation of the fractures using distal tibia fracture fixation implants (Depuy Synthes Inc. West Chester, PA) will be performed through standard approaches as judged by the operating surgeon. The implants can include, but is not limited to: 3.5 mm LCP Low Bend Medial Distal Tibia Plates, 3.5 mm LCP Antero-lateral Distal Tibia Plates, 3.5 mm LCP Posterior Distal Tibia Plates, or 2.7 mm / 3.5 mm LCP Distal Fibula Plates.

   4.2 Treatment Group: Enhanced Pre-Operative Planning In the treatment group, 20 patients randomized to enhanced pre-operative planning will include a 3D prototype of the distal tibia, fibula and talus-in addition to standard of care imaging (plain films 3 view, CT scans with sagittal, coronal and 3D reformations). On the injured extremity, discrete bone fragments are segmented and models of the study injury will then be imported into a computer aided design (CAD) software Unigraphics NX8 (Siemens PLM, Plano, TX). CAD models of the injured ankle will be converted into plastic prototypes using a Ultimaker 3D printer (Ultimaker B.V., Geldermalsen, Netherlands). Surgeons will use the 3D plastic prototype model to understand the geometry, displacement, and ideal reduced location of the fragments. Based on the addition of the 3D plastic prototype model, a second pre-operative plan will be documented. This will be compared to the initial pre-op plan to determine if the addition of the 3D prototype changed the surgeon's plan. The 3D plastic prototypes may be brought to the operating room (in the unsterile field) for reference during surgery as the surgeons execute the surgical plan. ORIF is then conducted to fix the fractures as per surgeon's standard of practice. The implants can include, but are not limited to: 3.5 mm LCP Low Bend Medial Distal Tibia Plates, 3.5 mm LCP Antero-lateral Distal Tibia Plates, 3.5 mm LCP Posterior Distal Tibia Plates, or 2.7 mm / 3.5 mm LCP Distal Fibula Plates (Depuy Synthes Inc. West Chester, PA).
5. Baseline and Follow-Up Assessments Demographics, mechanism of injury, and fracture classification will be collected at baseline. Patients will be followed over a 12-month period at 6 weeks, 26 weeks, and 52 weeks postoperatively. The outcome parameters being collected during the follow-up visits include re-operation, malunion and nonunion, other complications, Olerud and Molander Score, Numeric Pain Rating Scale (NPRS) for pain, and General Health Status. Radiographs as part of standard of care will be obtained of the anterior, lateral and oblique planes (3 views) to assess healing. The Schedule of Events details the requirements and procedures for each visit. Paper Case Report Forms (CRFs) will be used to document each follow-up assessment (as source documentation) and will then be entered electronically (eCRF) into an electronic data capture system. In cases when patients are not able to come in person for a follow-up assessment and all efforts to bring the patient in for an appointment have been exhausted, the option to complete the follow-up via telephone interview may be completed.

   5.1 Outcome Surveys Three outcome surveys will be obtained at each follow-up visit: 1) Olerud and Molander Scoring of Symptoms after Ankle Fracture, 2) Numeric Pain Rating Scale, and 3) General Health. The estimated total time to complete these three outcome surveys is 5 minutes.

   The Olerud and Molander Scoring of Symptoms after Ankle Fracture is a 9-question self-assessment of pain, stiffness, swelling, ability to climb stairs, run, jump, squat, use of supports, and work/activities of daily life. A total score out of 100 is calculated, with 100 equaling best or completely unimpaired. The Olerud and Molander Scoring of Symptoms after Ankle Fracture has been supported as a valid instrument, significantly correlating to a linear analog scale used to subjectively assess ankle function, range of motion in loaded dorsal extension, presence of osteoarthritis and presence of dislocation on radiographs. The Olerud and Molander Score also can capture minor subjective differences in disability and has a high correlation in test-retest reliability.

   A Numeric Pain Rating Scale (NPRS) (11-point numeric scale), a numeric version of the Visual Analog Scale for pain, will be used to assess the subject's current pain level. The NPRS is a 10 cm horizontal line, separated by 1cm integer increments, anchored with 0 = No Pain and 10 = Worst Possible Pain. The Numeric Rating Scale has been demonstrated to be valid in terms of construct validity, when compared to 5 other pain intensity measures such as Visual Analog Scale and Verbal Rating Scales. Subjects will be given this rating scale, self-administered, to record the number that best reflects their current pain. The NPRS takes less than 1 minute to complete. The NPRS can also be administered verbally by telephone.

   The subject's general health state will be measured using the Centers for Disease Control and Prevention's Health-Related Quality of Life, Healthy Days Core Module Question 1. This general health question is part of 4 items in the Healthy Days Core Module, which can be found in several national surveys, including the Behavioral Risk Factor Surveillance System and Medicare Health Outcome Survey. The validity of the CDC's HRQOL has been demonstrated.
6. Statistical Analysis The statistical analysis will be conducted using SPSS (IBM, version 18.0) and statistical significance set at p < α= .05 (two-tailed). Descriptive statistics will include frequency and percentages, as well as Chi-square analysis or Fisher's exact test (for cell sizes less than 5), to compare any differences at baseline between the two treatment groups. Any differences found at baseline, will be controlled for in the analysis as a covariate/confounding. The percentage of complications, such as infection, re-operation, malunion, and nonunion, within the two treatment groups will also be analyzed.

When comparing differences between the SOC versus enhanced pre-operative planning group (independent variable) and the Olerud and Molander Score and NPRS (ratio scales), both outcome/dependent variables capture pain. Therefore, a preliminary analysis of the correlation between these two dependent variables will be first assessed to determine appropriateness to use a multivariate analysis of variance (MANOVA), vs. two separate independent t-tests (Bonferroni correction α= .05/2). When comparing differences between the SOC versus enhanced pre-operative planning group with the categorical variable of general health, a Chi-square analysis or Fisher's exact test will be conducted.

The percentage of agreement between the pre and post-randomization pre-operative plan will be calculated and presented as a descriptive statistic. The number of items in agreement will be divided by the total number of items answered.

ELIGIBILITY:
Inclusion Criteria

1. Adults 18 to 75 years old.
2. Diagnosis of a closed or open, isolated intra-articular comminuted distal tibia fracture (OTA 43-C), with plans for delayed definitive surgery. May have concomitant fracture or injury of fibula.
3. Standard of care imaging available for pre-operative assessment and modeling
4. English speaking.
5. Available for follow-up for 12 months.
6. Patient signs informed consent.

Exclusion Criteria

1. History of musculoskeletal disease of the foot and/or ankle (i.e. arthritis).
2. Non-ambulatory prior to injury.
3. Bilateral lower extremity fractures.
4. Fracture of ipsilateral talus or calcaneus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome of Pain | Week 6 to week 52
  Patients will self-report pain using a numeric pain rating scale (NPRS), 11-point numeric scale. 0 = No pain and 10 = Worst Possible Pain
Patient Reported General Health State | Week 6 to week 52
  General Health State will be measured using the CDC HRQOL question 1, categorized into excellent, very good, good, fair, and poor.
Patient Functional Health Score | Week 6 to week 52
  Olerud and Molander Scoring System is a 9 question self-assessment of pain, stiffness, swelling, ability to climb stairs, run, jump, squat, use of supports, and work/activities of daily life. A total score of 100 is calculated, with 100 equaling best.

SECONDARY OUTCOMES:
Percentage of Agreement: Pre vs. Post Randomization Pre-Operative Plan | 0-1 mo
  Items on the pre and post randomization, pre-operative plan will be compared for agreement and presented as a descriptive statistic. The number of items in agreement will be divided by the total number of items answered, multiplied by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Hymes, M.D., Principal Investigator — Inova Fairfax Medical Campus
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will publish results through conferences and journals; de-identified group data results.

REFERENCES:
- [Background] Muller ME, Nazarian S, Koch P, Schatzker J. The comprehensive classification of fractures of long bones. Berlin: Springer; 1990.
- [Background] Topliss CJ, Jackson M, Atkins RM. Anatomy of pilon fractures of the distal tibia. J Bone Joint Surg Br. 2005 May;87(5):692-7. doi: 10.1302/0301-620X.87B5.15982. PMID 15855374
- [Background] Koulouvaris P, Stafylas K, Mitsionis G, Vekris M, Mavrodontidis A, Xenakis T. Long-term results of various therapy concepts in severe pilon fractures. Arch Orthop Trauma Surg. 2007 Jul;127(5):313-20. doi: 10.1007/s00402-007-0306-y. Epub 2007 Mar 13. PMID 17354011
- [Background] Pollak AN, McCarthy ML, Bess RS, Agel J, Swiontkowski MF. Outcomes after treatment of high-energy tibial plafond fractures. J Bone Joint Surg Am. 2003 Oct;85(10):1893-900. doi: 10.2106/00004623-200310000-00005. PMID 14563795
- [Background] Sands A, Grujic L, Byck DC, Agel J, Benirschke S, Swiontkowski MF. Clinical and functional outcomes of internal fixation of displaced pilon fractures. Clin Orthop Relat Res. 1998 Feb;(347):131-7. PMID 9520883
- [Background] Olerud C, Molander H. A scoring scale for symptom evaluation after ankle fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):190-4. doi: 10.1007/BF00435553. PMID 6437370
- [Background] Olerud and Molander Scoring System. J Orthop Trauma. 2006; 20: S102.
- [Background] Nilsson G, Jonsson K, Ekdahl C, Eneroth M. Outcome and quality of life after surgically treated ankle fractures in patients 65 years or older. BMC Musculoskelet Disord. 2007 Dec 20;8:127. doi: 10.1186/1471-2474-8-127. PMID 18096062
- [Background] Nilsson GM, Eneroth M, Ekdahl CS. The Swedish version of OMAS is a reliable and valid outcome measure for patients with ankle fractures. BMC Musculoskelet Disord. 2013 Mar 25;14:109. doi: 10.1186/1471-2474-14-109. PMID 23522388
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Newschaffer CJ. Validation of Behavioral Risk Factor Surveillance System (BRFSS) HRQOL measures in a statewide sample. Atlanta: U.S. Department of Health and Human Services, Public Health Service, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, 1998.